CLINICAL TRIAL: NCT03829709
Title: Electromiography Study in the Respiratory Muscle Training in Human Lymphotropic Virus Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, Phd, Director of Human Movement Department, Universidade Metodista de Piracicaba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2,629,073
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: HTLV-I Infections
MeSH Terms: conditions — HTLV-I Infections | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Rehabilitation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): The inspiratory muscle training (IMT) will be performed in the morning shift for 30 minutes, 3 times a week for 5 weeks. The first training session each week will be held at the LAERF under the direct supervision of the investigator and the other two home-based training sessions under the supervisor's distance supervision. They will receive the Threshold® IMT linear loading device, and guidelines for handling, posture and asepsis. The initial training load for each participant will be adjusted to 25% of PiMáx. Participants will be trained and instructed to do the exercise program on their own at home. Once a week, during the return to the laboratory the researcher will determine the new values for load (1st week 25%, 2nd week 35%, 3rd week 40%, 4th week 45%, 5th week 50%).
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — The first training session each week will be held at the LAERF under the direct supervision of the investigator and the other two home-based training sessions under the supervisor's distance supervision. They will receive the Threshold® IMT linear loading device, and guidelines for handling, posture and asepsis. The initial training load for each participant will be adjusted to 25% of PiMáx. Participants will be trained and instructed to do the exercise program on their own at home. Once a week, during the return to the laboratory the researcher will determine the new values for load (1st week 25%, 2nd week 35%, 3rd week 40%, 4th week 45%, 5th week 50%).

SUMMARY:
The main objective of the research will be to analyze, through surface electromyography, the impact of inspiratory muscle training before a supervised home training protocol in patients with human T-cell lymphotropic virus type 1 (HTLV-1). For this, a clinical, longitudinal, prospective, quantitative and single center trial will be carried out, aiming at home inspiratory muscle training lasting 5 weeks, 3 times a week, 30 minutes daily through the IMT Threshold, with 14 volunteers enrolled in the Laboratory of Studies in Functional Rehabilitation (LAERF) of the Federal University of Pará (UFPA). They will be classified as the manifestation of Tropical Spastic Paraparesis / Myelopathy (PET / MAH) for GP (PET / MAH probable) and GD (PET / MAH definitive) groups, obeying inclusion criteria. For characterization of expiratory flow rates and flows, as well as respiratory muscle strength, they will be submitted to spirometry and manovacuometry, pre, per, and post treatment, respectively. For the analysis of the electromyographic activity, the diaphragm, parasternal and sternocleidomastoid muscles will be counted in the follow-up during the analysis of inspiratory muscle strength, as well as once a week during the conduction of the inspiratory muscle training protocol. The collected data will be stored in a Microsoft Office Excel® 2010 worksheet and then submitted to statistical analysis using the Bioestat 5.0® program, adopting a standard error of 5%. The theoretical support of the research will have a bibliographical survey of scientific articles collected during the design of the project, and the accomplishment of the research. It is expected to map, through the surface electromyographic study, the impact of respiratory muscle training at a distance on the inspiratory muscle strength of patients with HTLV-I virus with probable or definitive PET / MAH.

DETAILED DESCRIPTION:
Human T-lymphotropic viruses, HTLV (Human Lymphotrophic Virus T), are retroviruses, which stand out as type 1 (HTLV-1) and type 2 (HTLV-2), the former being the etiologic agent of serious organ diseases such as leukemia adult T-cell lymphoma (ATLL), a neurological disorder, Tropical Spastic Paraparesis / HTLV-I-associated myelopathy (PET / HAM) and other non-malignant ophthalmologic, dermatological, rheumatic and osteomyelitis non-malignant disorders. For HTLV-2 it has not yet separated with some disease.

The highest prevalence of virus is found in countries of the Caribbean, South America, Melanesia Islands, West Africa and Japan. Brazil is an endemic country for infection and prevalence varies from state to state, being highest in Bahia, Pernambuco and Pará. The form of sexual transmission, hematologic for blood transfusions or accompanied by contaminated needles, mother-to-child verticalization, the passage of the lymphocyte infected by breast milk and also in the perinatal period.

The mechanism of the disease comes from the infection of several types of cells, such as T and B lymphocytes, monocytes and fibroblasts. However, its tropism is by TCD4 + cells. The form of contamination is cell-cell, thus being transferred from infected material to uninfected cells, modifying the immune system, as well as cell cells.

The main characteristic of HTLV infection is that in most cases the virus persists asymptomatic and undetectable by the immune system per year or until death in about 98% of the patients, while the hosts are able to transmit the virus. There are still no basic surveys on how severe forms of symptoms of graves occur in those infected.

In this context, when the individual becomes symptomatic, he is affected by chronic infection that may be associated with disabling diseases that compromise quality of life, such as the neurological disease PET-MAH. The onset is insidious with frequent changes in gait and urinary symptoms, mainly affecting the lower limbs such as spasticity, hyperreflexia, sensory-motor dysfunctions such as neuropathic or nociceptive pain, paresis, paralysis and paresthesia, urinary bladder disorders, muscle weakness and low back pain. The early diagnosis of motor complications in the face of the onset of neurological disease also contributes to the prevention of the installation of motor sensory sequelae if the physiotherapeutic treatment is established early. According to this reference, one of the aspects of preventive care refers to the functional autonomy correlated with physical conditioning in order to increase the strength and / or endurance of the skeletal muscles.

In this way, the possibility of morphological and functional changes in the respiratory system is also highlighted. With preventive therapeutic possibilities, the respiratory muscle training (TMR) appears to this indicator with reference to the maximum inspiratory and expiratory pressures (PiMáx and PeMáx). This procedure directly reflects on the patient's functionality, having as guideline the conduction of training protocols. The protocol should be conducted at least three days weekly frequently twice daily.

One tool to evaluate muscular behavior during TMR is surface electromyography (EMGs), which consists of a non-invasive detection of the muscular electrical activity by which it is presented graphically. It is constituted by the transcription of the sum of the electrical activity of all the active muscle fibers, through the positioning of electrodes on the skin. Thus, in order to verify the muscular activity of the respiratory dynamics related to inspiration, the main groups are the diaphragm, parasternal intercostal, sternocleidomastoid, abdominal rectus.

Therefore, the training requires time, availability and greater displacement of the patient to the outpatient treatment units, thus causing difficulties in adherence to the proposed therapy. To that end, it has been proposed ways that facilitate such conduction, such as home treatments, which, in most cases, the patient is supervised by the physiotherapist at least once a week presently followed by distance monitoring.

ELIGIBILITY:
Inclusion Criteria:

* volunteers of both sexes
* HTLV-1 positive serology with definitive or probable PET / MAH

Exclusion Criteria:

* pulmonary diseases
* serious comorbidities such as heart disease and uncontrolled arterial hypertension
* cognitive alterations that impede the conduction of the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Inspiratory and expiratory muscle force | Five weeks
  The evaluation of respiratory muscle strength will be performed by measuring the maximal inspiratory pressure (PiMáx) and expiratory (PeMAx) measurements with manovacuometer (+ - 300cmH2O). In order to perform the measurement of PiMáx and PeMáx, referring to inspiratory and expiratory muscle strength respectively. The values can range from 0 to 300 cmH2O, being 0 no strength and 300 maximum respiratory muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: João S Oliveira, phd, Study Chair — Universidade Metodista de Piracicaba
Locations (1):
- Universidade da Amazônia, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Magno Falcao LF, Falcao ASC, Medeiros Sousa RC, Vieira WB, de Oliveira RTM, Normando VMF, Dias GADS, Santos MCS, Rocha RSB, Yoshikawa GT, Koyama RVL, Fujihara S, Correa VAC, Fuzii HT, Quaresma JAS. CT Chest and pulmonary functional changes in patients with HTLV-associated myelopathy in the Eastern Brazilian Amazon. PLoS One. 2017 Nov 2;12(11):e0186055. doi: 10.1371/journal.pone.0186055. eCollection 2017. PMID 29095831
- [Result] Levy J, Prigent H, Bensmail D. Respiratory rehabilitation in multiple sclerosis: A narrative review of rehabilitation techniques. Ann Phys Rehabil Med. 2018 Jan;61(1):38-45. doi: 10.1016/j.rehab.2017.06.002. Epub 2017 Nov 8. PMID 29128525
- [Result] Nakamura T. HTLV-I-associated myelopathy/tropical spastic paraparesis (HAM/TSP): the role of HTLV-I-infected Th1 cells in the pathogenesis, and therapeutic strategy. Folia Neuropathol. 2009;47(2):182-94. PMID 19618340
- [Result] Nikoletou D, Man WD, Mustfa N, Moore J, Rafferty G, Grant RL, Johnson L, Moxham J. Evaluation of the effectiveness of a home-based inspiratory muscle training programme in patients with chronic obstructive pulmonary disease using multiple inspiratory muscle tests. Disabil Rehabil. 2016;38(3):250-9. doi: 10.3109/09638288.2015.1036171. Epub 2015 Apr 17. PMID 25885668
- [Result] Sa KN, Macedo MC, Andrade RP, Mendes SD, Martins JV, Baptista AF. Physiotherapy for human T-lymphotropic virus 1-associated myelopathy: review of the literature and future perspectives. J Multidiscip Healthc. 2015 Feb 23;8:117-25. doi: 10.2147/JMDH.S71978. eCollection 2015. PMID 25759588